CLINICAL TRIAL: NCT01524380
Title: A Double-blind and Randomized Trial of Ginkgo Biloba Extract Added to Risperidone in Treatment-naive First-episode Schizophrenia
Brief Title: Ginkgo Biloba Extract for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, co-Director, Psychiatric Research Center, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sch-FEP-001
Record Dates: First submitted 2012-01-28; First posted 2012-02-02 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; clinical trial; risperidone; ginkgo biloba extract; antioxidant
MeSH Terms: conditions — Schizophrenia | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginkgo biloba extract, antioxidant (Active Comparator): Active treatment with Ginkgo biloba extract
  Interventions: Drug: Ginkgo biloba extract
- Placebo (Placebo Comparator): Treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginkgo biloba extract — 400mg/day, twice a day, 10 weeks
  Other Names: EGb761
  Arms: Ginkgo biloba extract, antioxidant
Drug: Placebo — twice a day, 10 weeks
  Other Names: EGb761
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled trial of ginkgo biloba extract (Egb-761) as an add-on therapy to risperidone compared to risperidone plus placebo in the treatment of 200 treatment-naive first-episode patients with schizophrenia. The study addresses an immune dysfunction hypothesis of schizophrenia.

DETAILED DESCRIPTION:
OBJECTIVE: There is evidence that an excessive free radical production or oxidative stress may be involved in the pathophysiology of patients with schizophrenia. The investigators hypothesize that antioxidant therapy by using an add-on agent together with a well-proven antipsychotic drug may have favorable effects on some schizophrenic patients.

METHODS:

1. Clinical Trial: This is a randomized, double-blind and parallel controlled trial in treatment-naive first-episode patients with schizophrenia. The study consists of a 1-week stabilization phase, followed by 10 weeks of double-blind treatment. The total trial duration is 11 weeks.
2. Medications: Eligible patients are randomly assigned to either capsulized EGb(240mg.day) or identically capsulized placebo addition to the risperidone (2-6mg/day) in a double-blind fashion.
3. Assessment Procedures:

3.1. Primary Outcome Variable-psychopathology: Assessment instruments include the Positive and Negative Syndrome Scale (PANSS), and the Clinical Global Impression (CGI). Patients are interviewed at screening, at baseline and at every two weeks.

3.2. Cognitive tests: A comprehensive battery of tests encompassing the cognitive domains of executive function, attention, memory, perception, and general intellect is administered twice at baseline and at the end of 10-week treatment by a trained psychologist. Scoring follows standardized procedures.

3.3. Side Effects: Parkinsonism is rated with the Simpson-Angus Scale for extrapyramidal side effects. The Abnormal Involuntary Movement Scale (AIMS) is chosen to assess tardive dyskinesia (TD) severity. All of the AIMS and Simpson-Angus Rating Scales are administered by the same investigator at baseline and at baseline, and at week 5 and at week 10.

3.4. Plasma Measures: Venous blood from forearm vein is collected from healthy controls and patients with schizophrenia between 7 and 9 a.m. following an overnight fast. Serum Plasma malondialdehyde (MDA) levels and superoxide dismutase (SOD), glutathione peroxidase (GSH-Px) and catalase (CAT) activities will be analyzed using established procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizophreniform disorder;
* Duration of symptoms not longer than 60 months;
* No prior treatment with antipsychotic medication or, if previously treated, a total lifetime usage of less than 14 days;
* Between 16 and 40 years of age; and
* Current psychotic symptoms of moderate severity.

Exclusion Criteria:

* A DSM-IV Axis I diagnosis other than schizophrenia or schizophreniform;
* Documented disease of the central nervous system that can interfere with the trial assessments including, but not limited to stroke, tumor, Parkinson's disease, Huntington's disease, seizure disorder, history of brain trauma resulting in significant impairment, chronic, infection;
* Acute, unstable and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension);
* A clinically significant ECG abnormality in the opinion of the investigator;
* Pregnant or breast-feeding female;
* Use of disallowed concomitant therapy;
* History of severe allergy or hypersensitivity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
PANSS | 11 weeks
  PANSS

SECONDARY OUTCOMES:
CGI | 11 weeks
Cognition | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Y Zhang, MD/PhD, Principal Investigator — Beijing HuiLongGuan Hospital
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, China

REFERENCES:
- [Result] Zhang XY, Zhou DF, Su JM, Zhang PY. The effect of extract of ginkgo biloba added to haloperidol on superoxide dismutase in inpatients with chronic schizophrenia. J Clin Psychopharmacol. 2001 Feb;21(1):85-8. doi: 10.1097/00004714-200102000-00015. PMID 11199954